CLINICAL TRIAL: NCT05104567
Title: A Phase 2 Non-randomized, Open-label, Multi-cohort, Multi-center Study Assessing the Clinical Benefit of SAR444245 (THOR-707) Combined With Other Anticancer Therapies for the Treatment of Participants With Advanced and Metastatic Gastrointestinal Cancer
Brief Title: A Study of SAR444245 Combined With Other Anticancer Therapies for the Treatment of Participants With Gastrointestinal Cancer (Master Protocol) (Pegathor Gastrointestinal 203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16902; U1111-1251-4981 (Registry Identifier: ICTRP); MK-3475-B78 (Other: Merck Sharp & Dohme LLC.); KEYNOTE-B78 (Other: Merck Sharp & Dohme LLC.); 2021-002181-41 (EudraCT Number)
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Oesophageal Squamous Cell Carcinoma; Gastric Cancer; Hepatocellular Carcinoma; Colorectal Cancer; Oesophageal Adenocarcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Stomach Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms; Adenocarcinoma Of Esophagus | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Cohort A: ESCC Post PD-1/PD-L1; SAR444245 24 mcg/kg + Pembrolizumab as 2/3L Therapy (Experimental): Participants with advanced unresectable or metastatic esophageal squamous cell carcinoma (ESCC), regardless of programmed cell death-ligand 1 (PD-L1) expression (any combined positive score [CPS]), who had received at least 1 but no more than 2 prior lines of treatment and had progressed after primary or secondary resistance to an anti-programmed cell death-1 (PD-1)/PD-L1 based regimen were included in this cohort. Participants received SAR444245 24 microgram per kilogram (mcg/kg) along with pembrolizumab 200 milligram (mg) via intravenous (IV) infusion every 3 weeks (q3w) on Day 1 of each cycle (each cycle is 21 days) (as second-line or third-line [2/3L] therapy), until disease progression (PD), unacceptable adverse event (AE) or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort B1: GC/GEJ PD-1/PD-L1 naïve non-MSI-H CPS >=1 (Experimental): Cohort B1: GC/GEJ PD-1/PD-L1 naïve non-MSI-H CPS >=1; SAR444245 24mcg/kg+Pembrolizumab as 1-3L Therapy. Participants with advanced unresectable or metastatic gastric cancer (GC) or Siewert Type 2 & 3 gastro-esophageal junction adenocarcinoma (GEJ) and for whom standard of care (SOC) was not in best interest or where no SOC was established, non-high-level microsatellite instability (MSI-H) disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS >=1 GC/GEJ were included in this cohort. Participants received SAR444245 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as first to [1-]3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort B2: GC/GEJ PD-1/PD-L1 naïve non-MSI-H CPS <1 (Experimental): Cohort B2: GC/GEJ PD-1/PD-L1 naïve non-MSI-H CPS <1; SAR444245 24 mcg/kg+Pembrolizumab as 1-3L Therapy. Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS <1 GC/GEJ were included in this cohort. Participants received SAR444245 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort B3: GC/GEJ Post PD-1/PD-L1 non-MSI-H; SAR444245 24 mcg/kg + Pembrolizumab as 2-4L Therapy (Experimental): Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had received atleast 1 and no more than 3 prior lines of treatment and had progressed after primary or secondary resistance to an anti-PD-1/PD-L1-based regimen (regardless of the disease CPS status) were included in this cohort. Participants received SAR444245 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2-fourth [4]L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort C: HCC Post PD-1/PD-L1; SAR444245 24 mcg/kg + Pembrolizumab as 2/3L Therapy (Experimental): Participants with advanced unresectable or metastatic hepatocellular carcinoma (HCC), regardless of any CPS, who relapsed on prior PD-1/PD-L1-based regimens, with at least stable disease (SD) as best response and with no more than 2 prior lines of treatment were included in this cohort. Participants received SAR444245 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort D1: CRC non-MSI-H any RAS; SAR444245 24 mcg/kg + Pembrolizumab as 3-6L Therapy (Experimental): Participants with advanced unresectable or metastatic colorectal cancer (CRC), regardless of any CPS, non-MSI-H disease, any RAS type, who had progressed on prior regimens having contained fluoropyrimidine, oxaliplatin, irinotecan, with either bevacizumab or cetuximab, and with no more than 5 prior lines of treatments were included in this cohort. Participants received SAR444245 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 3-sixth [6]L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort D2: CRC non-MSI-H RAS Wild Type; SAR444245 24 mcg/kg + Cetuximab as 3-6L Therapy (Experimental): Participants with advanced unresectable or metastatic CRC, regardless of any CPS, non-MSI-H disease, RAS wild type, who had progressed on prior regimens having contained fluoropyrimidine, oxaliplatin, irinotecan, with either bevacizumab or cetuximab, and with no more than 5 prior lines of treatments were included in this cohort. Participants received SAR444245 24 mcg/kg q3w on Day 1 of each cycle along with cetuximab as an initial loading dose of 400 mg/square meter (m^2) on Cycle 1 Day 1 followed by 250 mg/m^2 starting via IV infusion once weekly from Cycle 1 Day 8 (each cycle is 21 days) (as 3-6L therapy) until PD.
  Interventions: Drug: THOR-707; Drug: Cetuximab

INTERVENTIONS:
Drug: THOR-707 — Solution for infusion: intravenous infusion
  Other Names: Pegenzileukin
Drug: Pembrolizumab — Solution for infusion: intravenous infusion
  Other Names: KEYTRUDA®
  Arms: Cohort A: ESCC Post PD-1/PD-L1; SAR444245 24 mcg/kg + Pembrolizumab as 2/3L Therapy; Cohort B1: GC/GEJ PD-1/PD-L1 naïve non-MSI-H CPS >=1; Cohort B2: GC/GEJ PD-1/PD-L1 naïve non-MSI-H CPS <1; Cohort B3: GC/GEJ Post PD-1/PD-L1 non-MSI-H; SAR444245 24 mcg/kg + Pembrolizumab as 2-4L Therapy; Cohort C: HCC Post PD-1/PD-L1; SAR444245 24 mcg/kg + Pembrolizumab as 2/3L Therapy; Cohort D1: CRC non-MSI-H any RAS; SAR444245 24 mcg/kg + Pembrolizumab as 3-6L Therapy
Drug: Cetuximab — Solution for infusion: intravenous infusion
  Other Names: ERBITUX®
  Arms: Cohort D2: CRC non-MSI-H RAS Wild Type; SAR444245 24 mcg/kg + Cetuximab as 3-6L Therapy

SUMMARY:
The study is a phase 2 non-randomized, open-label, multi-cohort, multi-center study assessing the clinical benefit of SAR444245 (THOR-707) combined with other anticancer therapies for the treatment of participants aged 18 years and older with advanced and metastatic gastrointestinal cancer. This study is structured as a master protocol for the investigation of SAR444245 with other anticancer therapies.

Sub study 01 - Cohort A aims to establish proof-of-concept that combining the non-alpha-IL2 SAR444245 with the anti-PD1 antibody pembrolizumab will result in a significant increase in the percentage of patients experiencing an objective response in the setting of advanced unresectable or metastatic esophageal squamous cell carcinoma (ESCC).

Sub study 02 - Cohort B1, B2 and B3 would focus on non MSI-H tumors with a large unmet need to establish proof-of-concept that combining the non-alpha-IL2 SAR444245 with the anti-PD1 antibody pembrolizumab will result in a significant increase in the percentage of patients experiencing an objective response in the setting of advanced unresectable or metastatic gastric cancer or gastro-esophageal junction adenocarcinoma (GC/GEJ), especially with low PD-L1 expression or after progression on prior PD1/PD-L1-based regimens.

Sub study 03 - Cohort C aims to establish proof-of-concept that combining the non-alpha-IL2 SAR444245 with the anti-PD1 antibody pembrolizumab will result in a significant increase in the percentage of patients experiencing an objective response in participants with advanced unresectable or metastatic HCC who relapsed on prior PD1/PD-L1-based regimens.

Sub study 04 - Cohort D1 and D2 aims to establish proof-of-concept that combining the non-alpha-IL2 SAR444245 with either the anti-PD1 antibody pembrolizumab or with the anti-EGFR IgG1 antibody cetuximab will result in a significant increase in the percentage of patients experiencing an objective response in the setting of advanced unresectable or metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
The duration of the study for an individual patient will start from the signature of the main informed consent and include a screening period of up to 28 days, a treatment period [max 35 cycles {cohort A; B1,B2, B3, C and D1} = 735 days or until PD {cohort D2}], an end-of-treatment visit at least 30 days following the last administration of study drug (or until the patient receives another anticancer therapy, whichever is earlier), and a follow-up visit 3 months after treatment discontinuation and every 3 months following, until disease progression, or initiation of another antitumor treatment, or death, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age (or country's legal age of majority if >18 years), at the time of signing the informed consent.
* Participants with:

  * Sub-study01: Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic esophageal cancer of the squamous cell carcinoma subtype.
  * Sub-study02: Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ.
  * Sub-study03: Histologically or cytologically confirmed diagnosis of advanced unresectable or metastatic hepatocellular carcinoma (HCC), or clinically by AASLD criteria in cirrhotic patients.
  * Sub-study04: Histologically or cytologically confirmed diagnosis of advanced unresectable or mCRC. Only patients with non-MSI-H disease are eligible.
* Participants (all sub-studies) must have at least one measurable lesion.
* Mandatory baseline biopsy for the first 20 participants to enroll in sub-study01, sub-study02 and sub-study04. On-treatment biopsy for at least 20 participants in sub-study04. On-treatment biopsies are otherwise optional per Investigator's discretion for the other cohorts.
* Females are eligible to participate if they are not pregnant or breastfeeding, not a woman of childbearing potential (WOCBP) or are a WOCBP that agrees:

  * to use approved contraception method and submit to regular pregnancy testing prior to treatment and for at least 120 days (for Cohort A, B1, B2, B3, C, and D1) or 60 days (for Cohort D2) [corresponding to the time needed to eliminate any study intervention(s)].
  * and to refrain from donating or cryopreserving eggs for 120 days after discontinuing study treatment.
* Males are eligible to participate if they agree to refrain from donating or cryopreserving sperm, and either abstain from heterosexual intercourse OR use approved contraception during study treatment and for at least 3 days [corresponding to time needed to eliminate SAR444245] after the last dose of SAR444245.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≥2.
* Poor organ function.
* Active brain metastases or leptomeningeal disease.
* History of allogenic or solid organ transplant.
* Last administration of prior antitumor therapy or any investigational treatment within 28 days or less than 5 times the half-life, whichever is shorter; major surgery within 28 days prior to first IMP administration.
* Comorbidity requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 2 weeks of IMP initiation. Inhaled or topical steroids are permitted, provided that they are not for treatment of an autoimmune disorder. Participants who require a brief course of steroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded).
* Antibiotic use (excluding topical antibiotics) ≤14 days prior to first dose of IMP.
* Severe or unstable cardiac condition within 6 months prior to starting study treatment.
* Active, known, or suspected autoimmune disease that has required systemic treatment in the past 2 years.
* Participants with baseline SpO2 ≤92% (without oxygen therapy). - Participant has received prior IL2-based anticancer treatment.
* Participants on sub-study02 cohort B1 and B2 or sub-study 04 - cohort D1 with prior treatment with an agent that blocks the PD-1/PD-L1 pathway.
* Receipt of a live-virus or live attenuated-virus vaccination within 28 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (3):
  - City of Hope Site Number : 8400007, Duarte, California
  - AdventHealth Orlando Site Number : 8400005, Orlando, Florida
  - Seattle Cancer Care Alliance Site Number : 8400009, Seattle, Washington
- Belgium (3):
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560003, Edegem
  - Investigational Site Number : 0560001, Leuven
- Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago, Chile
- Investigational Site Number : 1560002, Wuhan, China
- France (5):
  - Investigational Site Number : 2500004, Bordeaux
  - Investigational Site Number : 2500006, Brest
  - Investigational Site Number : 2500002, Paris
  - Investigational Site Number : 2500005, Poitiers
  - Investigational Site Number : 2500001, Villejuif
- Italy (3):
  - Investigational Site Number : 3800001, Rozzano, Lombardy
  - Investigational Site Number : 3800003, Milan
  - Investigational Site Number : 3800002, Milan
- Netherlands (2):
  - Investigational Site Number : 5280001, Amsterdam
  - Investigational Site Number : 5280003, Rotterdam
- South Korea (4):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
- Spain (7):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Santander, Cantabria
  - Investigational Site Number : 7240101, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240003, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240001, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16902 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25203&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 29 centers (corresponds to number of site which screened at least one participant) in 9 countries. Out of 193 participants who were screened from 09 December 2021 to 26 October 2022, a total of 138 participants were enrolled in the study and were assigned to 1 of the 7 cohorts (Cohorts A, B1, B2, B3, C, D1 and D2) based on their disease type.
Pre-assignment Details: Note: Reason for not completed = Reason for permanent full intervention discontinuation.
Groups:
- Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy: Participants with advanced unresectable or metastatic esophageal squamous cell carcinoma (ESCC), regardless of programmed cell death-ligand 1 (PD-L1) expression (any combined positive score [CPS]), who had received at least 1 but no more than 2 prior lines of treatment and had progressed after primary or secondary resistance to an anti-programmed cell death-1 (PD-1)/PD-L1 based regimen were included in this cohort. Participants received pegenzileukin 24 microgram per kilogram (mcg/kg) along with pembrolizumab 200 milligram (mg) via intravenous (IV) infusion every 3 weeks (q3w) on Day 1 of each cycle (each cycle is 21 days) (as second-line or third-line [2/3L] therapy), until disease progression (PD), unacceptable adverse event (AE) or other full permanent discontinuation criteria was met or completion of Cycle 35.
- CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy: Participants with advanced unresectable or metastatic gastric cancer (GC) or Siewert Type 2 & 3 gastro-esophageal junction adenocarcinoma (GEJ) and for whom standard of care (SOC) was not in best interest or where no SOC was established, non-high-level microsatellite instability (MSI-H) disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS >=1 GC/GEJ were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as first to [1-]3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS <1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy: Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS <1 GC/GEJ were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy: Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had received atleast 1 and no more than 3 prior lines of treatment and had progressed after primary or secondary resistance to an anti-PD-1/PD-L1-based regimen (regardless of the disease CPS status) were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2-fourth [4]L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy: Participants with advanced unresectable or metastatic hepatocellular carcinoma (HCC), regardless of any CPS, who relapsed on prior PD-1/PD-L1-based regimens, with at least stable disease (SD) as best response and with no more than 2 prior lines of treatment were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy: Participants with advanced unresectable or metastatic colorectal cancer (CRC), regardless of any CPS, non-MSI-H disease, any RAS type, who had progressed on prior regimens having contained fluoropyrimidine, oxaliplatin, irinotecan, with either bevacizumab or cetuximab, and with no more than 5 prior lines of treatments were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 3-sixth [6]L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy: Participants with advanced unresectable or metastatic CRC, regardless of any CPS, non-MSI-H disease, RAS wild type, who had progressed on prior regimens having contained fluoropyrimidine, oxaliplatin, irinotecan, with either bevacizumab or cetuximab, and with no more than 5 prior lines of treatments were included in this cohort. Participants received pegenzileukin 24 mcg/kg q3w on Day 1 of each cycle along with cetuximab as an initial loading dose of 400 mg/square meter (m^2) on Cycle 1 Day 1 followed by 250 mg/m^2 starting via IV infusion once weekly from Cycle 1 Day 8 (each cycle is 21 days) (as 3-6L therapy) until PD.
Period: Overall Study
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS <1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Started | 5 | 22 | 19 | 18 | 20 | 30 | 24
Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 21 | 19 | 18 | 20 | 30 | 24
Not completed — Adverse event: Related to Coronavirus Disease 2019 (COVID-19) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event: Not related to COVID-19 | 0 | 5 | 3 | 1 | 3 | 2 | 0
Not completed — Progressive disease | 3 | 13 | 13 | 17 | 17 | 28 | 24
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The exposed population included all participants who had given their informed consent and received at least one dose of study treatment (pegenzileukin or other anticancer therapies).
Groups:
- Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy: Participants with advanced unresectable or metastatic ESCC, regardless of PD-L1 expression (any CPS), who had received at least 1 but no more than 2 prior lines of treatment and had progressed after primary or secondary resistance to an anti-PD-1/PD-L1 based regimen were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy: Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS >=1 GC/GEJ were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy: Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS <1 GC/GEJ were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy: Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had received atleast 1 and no more than 3 prior lines of treatment and had progressed after primary or secondary resistance to an anti-PD-1/PD-L1-based regimen (regardless of the disease CPS status) were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2-4L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy: Participants with advanced unresectable or metastatic HCC, regardless of any CPS, who relapsed on prior PD-1/PD-L1-based regimens, with at least SD as best response and with no more than 2 prior lines of treatment were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy: Participants with advanced unresectable or metastatic CRC, regardless of any CPS, non-MSI-H disease, any RAS type, who had progressed on prior regimens having contained fluoropyrimidine, oxaliplatin, irinotecan, with either bevacizumab or cetuximab, and with no more than 5 prior lines of treatments were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 3-6L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy: Participants with advanced unresectable or metastatic CRC, regardless of any CPS, non-MSI-H disease, RAS wild type, who had progressed on prior regimens having contained fluoropyrimidine, oxaliplatin, irinotecan, with either bevacizumab or cetuximab, and with no more than 5 prior lines of treatments were included in this cohort. Participants received pegenzileukin 24 mcg/kg q3w on Day 1 of each cycle along with cetuximab as an initial loading dose of 400 mg/m^2 on Cycle 1 Day 1 followed by 250 mg/m^2 starting via IV infusion once weekly from Cycle 1 Day 8 (each cycle is 21 days) (as 3-6L therapy) until PD.
- Total: Total of all reporting groups
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy | Total
Number analyzed (Participants) | 5 | 22 | 19 | 18 | 20 | 30 | 24 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (4.4) | 58.1 (10.3) | 56.5 (13.1) | 58.3 (10.9) | 65.7 (8.8) | 62.7 (12.1) | 61.7 (10.0) | 60.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7 | 4 | 6 | 11 | 7 | 42
  Male | 3 | 17 | 12 | 14 | 14 | 19 | 17 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 2 | 6 | 3 | 0 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 13 | 15 | 10 | 14 | 30 | 18 | 103
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 8 | 2 | 1 | 3 | 0 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 millimeter (mm) (<1 centimeter [cm]). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 8 months
Population: The efficacy population included all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 5
percentage of participants | 20.0 [1.0 to 65.7]

2. Primary Outcome: Cohorts B1, B2 and B3: Objective Response Rate
Description: ORR was defined as the percentage of participants who had a confirmed CR or PR as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 25 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy: Participants with advanced unresectable or metastatic GC or Siewert Type 2 & 3 GEJ and for whom SOC was not in best interest or where no SOC was established, non-MSI-H disease and had not received more than 2 prior lines of treatment that did not include an anti-PD-1/PD-L1-based regimen with the level of PD-L1 expression at baseline as CPS <1 GC/GEJ were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 1-3L therapy), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
Arm/Group | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy
Number analyzed (Participants) | 22 | 19 | 18
percentage of participants | 13.6 [3.8 to 31.6] | 5.3 [0.3 to 22.6] | 11.1 [2.0 to 31.0]

3. Primary Outcome: Cohort C: Objective Response Rate
Description: as for outcome 2
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 20 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 20
percentage of participants | 5.0 [0.3 to 21.6]

4. Primary Outcome: Cohorts D1 and D2: Objective Response Rate
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 30 | 24
percentage of participants | 0 [0.0 to 9.5] | 8.3 [1.5 to 24.0]

5. Secondary Outcome: All Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened (according to the Investigator's opinion) or became serious during the TE period.
Time Frame: From first dose of study treatment administration (Day 1) up to 30 days post last dose of study treatment administration, up to approximately 9 months (Cohorts A, D1 and D2), 26 months (Cohorts B1, B2 and B3) and 21 months (Cohort C)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 5 | 22 | 19 | 18 | 20 | 30 | 24
Participants
  TEAEs | 5 | 22 | 19 | 18 | 19 | 30 | 24
  TESAEs | 2 | 17 | 13 | 9 | 7 | 19 | 11

6. Secondary Outcome: All Cohorts: Time to Response (TTR)
Description: TTR was defined as the time from the date of first study treatment administration to the first tumor assessment at which the overall response was recorded as PR or CR that was subsequently confirmed as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 8 months (Cohort A, D1 and D2), 25 months (Cohort B1, B2 and B3), 20 months (Cohort C)
Population: The efficacy population included all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment. Only participants with confirmed CR or PR were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 1 | 3 | 1 | 2 | 1 | 0 | 2
months | 1.9 (NA) — NA indicates that the standard deviation (SD) was not estimable for 1 participant. | 2.1 (0.2) | 4.2 (NA) — NA indicates that the SD was not estimable for 1 participant. | 3.0 (1.3) | 6.0 (NA) — NA indicates that the SD was not estimable for 1 participant. |  | 2.0 (0.1)

7. Secondary Outcome: All Cohorts: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first tumor assessment at which the overall response was recorded as CR or PR that was subsequently confirmed to the date of first documentation of objective PD before the initiation of any post-treatment anti-cancer therapy or death due to any cause, whichever occurred first, as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 1 | 3 | 1 | 2 | 1 | 0 | 2
months | NA [NA to NA] — NA indicates that the median, upper and lower limit of 90% confidence interval (CI) were not estimable due to insufficient number of participants with events. | 13.1 [NA to NA] — NA indicates that the upper and lower limit of 90% CI were not estimable, as there were insufficient numbers of participants with 2/3 participants censored prior to any event. | NA [NA to NA] — NA indicates that the median, upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. | 8.8 [8.6 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — NA indicates that the median, upper and lower limit of 90% CI were not estimable due to insufficient number of participants with events. |  | 4.1 [4.1 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events.

8. Secondary Outcome: All Cohorts: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with clinical benefit (confirmed CR or PR as best overall response [BOR], or SD lasting at least 6 months), as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. BOR was defined as the best response recorded from the start of the study treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 5 | 22 | 19 | 18 | 20 | 30 | 24
percentage of participants | 40.0 [7.6 to 81.1] | 22.7 [9.4 to 42.0] | 10.5 [1.9 to 29.6] | 11.1 [2.0 to 31.0] | 10.0 [1.8 to 28.3] | 6.7 [1.2 to 19.5] | 12.5 [3.5 to 29.2]

9. Secondary Outcome: All Cohorts: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first study treatment to the date of the first documentation of objective PD or death due to any cause, whichever occurred first, as per RECIST v 1.1. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 5 | 22 | 19 | 18 | 20 | 30 | 24
months | NA [2.2 to NA] — NA indicates that the median and upper limit of 90% CI were not estimable due to insufficient number of participants with events. | 1.9 [1.2 to 2.9] | 2.0 [1.4 to 3.5] | 2.1 [1.8 to 2.2] | 2.1 [1.9 to 2.2] | 2.0 [1.9 to 2.1] | 2.1 [2.0 to 4.1]

10. Secondary Outcome: Maximum Concentration Observed (Cmax) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of Cmax of pegenzileukin. The pharmacokinetic (PK) parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: The PK population included all participants from exposed population with at least one PK concentration available after the first dose of study treatment. Same dose of pegenzileukin was administered to all participants in Cohorts A, B1, B2, B3, C, D1 and D2 of the study. Hence PK analysis was combined for all the cohorts. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- All Cohorts: Pegenzileukin 24 mcg/kg: All participants received pegenzileukin 24 mcg/kg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days), until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 35
nanograms per milliliter (ng/mL)
  Day 1 Cycle 1 | 417 (109)
  Day 1 Cycle 4: number analyzed (Participants) | 12
  Day 1 Cycle 4 | 369 (118)

11. Secondary Outcome: Last Concentration Observed Above the Lower Limit of Quantification (Clast) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of Clast of pegenzileukin. The PK parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 35
ng/mL
  Day 1 Cycle 1 | 17.6 (13.4)
  Day 1 Cycle 4: number analyzed (Participants) | 9
  Day 1 Cycle 4 | 13.0 (6.11)

12. Secondary Outcome: Time of the Last Concentration Observed Above the Lower Limit of Quantification (Tlast) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of tlast of pegenzileukin. The PK parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 35
Hours (h)
  Day 1 Cycle 1 | 69.45 [43.00 to 76.77]
  Day 1 Cycle 4: number analyzed (Participants) | 9
  Day 1 Cycle 4 | 68.82 [46.28 to 72.58]

13. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated Using the Trapezoidal Method From Time Zero to Tlast (AUClast) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of AUClast of pegenzileukin. The PK parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 35
ng*h/mL
  Day 1 Cycle 1 | 8940 (1930)
  Day 1 Cycle 4: number analyzed (Participants) | 9
  Day 1 Cycle 4 | 7100 (2330)

14. Secondary Outcome: Area Under the Concentration Versus Time Curve Extrapolated to Infinity (AUC) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of AUC of pegenzileukin. The PK parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 34
ng*h/mL
  Day 1 Cycle 1 | 9270 (1990)
  Day 1 Cycle 4: number analyzed (Participants) | 9
  Day 1 Cycle 4 | 7330 (2340)

15. Secondary Outcome: Observed Accumulation Ratio (Rac) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of Rac of pegenzileukin. Rac was calculated as AUC at Cycle 4 Day 1/AUC at Cycle 1 Day 1. The PK parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 9
ratio | 0.772 (0.150)

16. Secondary Outcome: Observed Accumulation Ratio Based on Cmax (Rac,Cmax) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of Rac,cmax of pegenzileukin. Rac,cmax was calculated as Cmax at Cycle 4 Day 1/Cmax at Cycle 1 Day 1. The PK parameters were calculated using non-compartmental method.
Time Frame: Day 1 Cycle 1 and Day 1 Cycle 4 (each cycle is 21 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Cohorts: Pegenzileukin 24 mcg/kg
Number analyzed (Participants) | 12
ratio | 0.887 (0.173)

17. Secondary Outcome: Cohort D2: Concentration Observed Just Before Intervention Administration During Repeated Dosing (Ctrough) of Cetuximab
Description: Blood samples were collected at specified timepoints for the assessment of Ctrough of Cetuximab. The PK parameters were calculated using non-compartmental method.
Time Frame: Cycles 1, 2, 3, 4, 6 and 8 (each cycle is 21 days)
Population: The PK population included all participants from exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 19
ng/mL
  Cycle 1: number analyzed (Participants) | 18
  Cycle 1 | 0.0 (0.0)
  Cycle 2 | 61689.5 (29031.6)
  Cycle 3: number analyzed (Participants) | 14
  Cycle 3 | 61647.1 (41623.9)
  Cycle 4: number analyzed (Participants) | 10
  Cycle 4 | 88670.0 (53487.3)
  Cycle 6: number analyzed (Participants) | 9
  Cycle 6 | 84377.8 (39150.0)
  Cycle 8: number analyzed (Participants) | 4
  Cycle 8 | 118375.0 (51770.9)

18. Secondary Outcome: Cohort D2: Concentration at End of Infusion (Ceoi) of Cetuximab
Description: Blood samples were collected at specified timepoints for the assessment of Ceoi of Cetuximab. The PK parameters were calculated using non-compartmental method.
Time Frame: Cycles 1, 2, 3, 4, 6 and 8 (each cycle is 21 days)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 18
ng/mL
  Cycle 1: number analyzed (Participants) | 17
  Cycle 1 | 245352.9 (57442.3)
  Cycle 2 | 209111.1 (52687.6)
  Cycle 3: number analyzed (Participants) | 14
  Cycle 3 | 214857.1 (69955.9)
  Cycle 4: number analyzed (Participants) | 10
  Cycle 4 | 236700.0 (63756.6)
  Cycle 6: number analyzed (Participants) | 9
  Cycle 6 | 233777.8 (53473.8)
  Cycle 8: number analyzed (Participants) | 4
  Cycle 8 | 248500.0 (59991.7)

19. Secondary Outcome: All Cohorts: Number of Participants With Anti-Drug Antibodies (ADAs) Against Pegenzileukin
Description: Blood samples were collected at specified timepoints to assess the presence of ADA against pegenzileukin. Treatment-emergent ADA was defined as at least one treatment-induced or treatment-boosted ADA. Treatment-induced ADA was defined as ADA that developed during the TE period and without pre-existing ADA (including participants without pre-treatment samples). Treatment-boosted ADA was defined as pre-existing ADA that was boosted during the TE period to a significant higher titer than the baseline. Number of participants with treatment-emergent ADA is presented.
Time Frame: as for outcome 5
Population: The ADA population included all participants from exposed population with at least one ADA result (positive, negative or inconclusive) after the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
Number analyzed (Participants) | 5 | 22 | 18 | 16 | 20 | 30 | 23
Participants | 1 | 2 | 5 | 0 | 3 | 11 | 3

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from first dose of study treatment administration (Day 1) up to 30 days post last dose of study treatment administration, up to approximately 9 months (Cohorts A, D1 and D2), 26 months (Cohorts B1, B2 and B3) and 21 months (Cohort C). All-cause mortality (deaths) were collected from first dose of study treatment administration (Day 1) to the end of follow-up for death for each participant, up to approximately 19 months.
Description: Analysis was performed on the exposed population.
Arm/Group | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy
All-Cause Mortality (participants affected / at risk) | 1/5 | 16/22 | 15/19 | 12/18 | 6/20 | 24/30 | 18/24
Serious Adverse Events (participants affected / at risk) | 2/5 | 17/22 | 13/19 | 9/18 | 7/20 | 19/30 | 11/24
Other Adverse Events (participants affected / at risk) | 5/5 | 20/22 | 18/19 | 17/18 | 19/20 | 30/30 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy (N=5) | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy (N=22) | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy (N=19) | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy (N=18) | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy (N=20) | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy (N=30) | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy (N=24)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (5) | 1 (3) | 1 (1) | 2 (4) | 4 (5) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure To Thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune Effector Cell-Associated Neurotoxicity Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Antral Vascular Ectasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Intestinal Pseudo-Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice Cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric Compression (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 2 (3)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: ESCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy (N=5) | CohortB1:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS>=1:Pegenzileukin24mcg/kg+Pembrolizumab as 1-3LTherapy (N=22) | CohortB2:GC/GEJ PD-1/PD-L1 naïve Non-MSI-H CPS<1:Pegenzileukin24 mcg/kg+Pembrolizumab as 1-3LTherapy (N=19) | Cohort B3: GC/GEJ Post PD-1/PD-L1 Non-MSI-H: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2-4L Therapy (N=18) | Cohort C: HCC Post PD-1/PD-L1: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy (N=20) | Cohort D1: CRC Non-MSI-H Any RAS: Pegenzileukin 24 mcg/kg + Pembrolizumab as 3-6L Therapy (N=30) | Cohort D2: CRC Non-MSI-H RAS Wild Type: Pegenzileukin 24 mcg/kg + Cetuximab as 3-6L Therapy (N=24)
Covid-19 (Infections and infestations) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 1 (1) | 3 (23) | 1 (1) | 3 (5) | 2 (2) | 4 (4) | 3 (9)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abnormal Loss Of Weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (6) | 10 (11) | 6 (6) | 3 (3) | 8 (9) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Mood Swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain Fog (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Hot Flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 5 (6) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Larynx Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 7 (8) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (5) | 3 (3) | 0 (0)
Angular Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 5 (7) | 3 (3) | 1 (1) | 6 (8) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 6 (12) | 7 (9) | 4 (4) | 5 (5) | 6 (8) | 7 (7)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (6) | 9 (10) | 6 (6) | 7 (7) | 11 (16) | 7 (8)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 4 (5) | 3 (4) | 2 (2) | 9 (14) | 5 (5)
Biliary Obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dermatitis Psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Hand Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 8 (8)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 1 (2) | 6 (6) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital Rubella Syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (4) | 11 (18) | 4 (5) | 7 (7) | 8 (12) | 16 (23) | 8 (12)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (4) | 6 (6) | 3 (3) | 3 (5) | 3 (3) | 5 (7)
Influenza Like Illness (General disorders) | 1 (1) | 4 (18) | 5 (27) | 5 (13) | 6 (10) | 17 (31) | 5 (18)
Localised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 3 (5) | 4 (6) | 5 (5) | 4 (4) | 5 (8) | 3 (3)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 4 (7) | 8 (9) | 6 (11) | 6 (12) | 13 (24) | 11 (14)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to early discontinuation based on strategic sponsor decision not driven by any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT05104567/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT05104567/SAP_001.pdf